CLINICAL TRIAL: NCT02088034
Title: Promotora-led Intervention to Promote Weight Loss in Latinas At-risk for Diabetes
Brief Title: Intervention to Promote Weight Loss in Latinas At-risk for Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21273
Record Dates: First submitted 2014-03-05; First posted 2014-03-14 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Promotora-led Intervention (Experimental): The Promotora-led Intervention consists of a core curriculum or 12 group sessions of 90 minute duration over a 12-week period and will be followed by a maintenance phase of 10 biweekly and then monthly 90-minute sessions during months 4 through 12. One promotora will lead each session in Spanish, exploring such topics as being active, low-fat diets, portion control, self monitoring, problem solving and life-style changes.
  Interventions: Behavioral: Promotora-led Intervention
- Usual care (Active Comparator): One physician visit at Puentes de Salud or Congreso Health Center to discuss healthy lifestyle behaviors that promote weight loss and diabetes prevention. During that visit, UC participants will also receive standard educational materials in Spanish from the NIDDK Weight-control Information Network covering the same topics. UC participants will receive another physician visit upon completion of 1-year follow-up to review laboratory assessments.
  Interventions: Other: Usual Care
- Metformin Therapy (Active Comparator): Participants randomized to the metformin arm of the study will receive this medication from months 1 through 12 after randomization. Subjects will receive 850 mg daily for 1 month and increase to 850 mg twice daily thereafter if no side effects are experienced.
  Interventions: Drug: Metformin Therapy

INTERVENTIONS:
Behavioral: Promotora-led Intervention — Behavioral life-style program lead by a team of trained community health workers (called promotoras) with 2 principal goals - encouraging participants to lose 7% of their total weight and complete 150 minutes of moderate physical activity per week.
  Other Names: ILI
  Arms: Promotora-led Intervention
Drug: Metformin Therapy — Participants in this group will receive metformin 850 mg bid for one year.
  Other Names: Metformin
  Arms: Metformin Therapy
Other: Usual Care — Participants in this arm will attend one physician visit to discuss healthy lifestyle behaviors and will receive standard educational materials.
  Other Names: Control
  Arms: Usual care

SUMMARY:
The overarching goal of this project is to develop and test a behavioral intervention delivered by promotoras to help at-risk Latinas lose weight and prevent diabetes.

DETAILED DESCRIPTION:
The goal of the proposed research is to compare two evidence-based strategies for preventing type 2 diabetes - promotora-led lifestyle intervention and metformin - vs. usual care (UC) among Latinas in a "real world" setting. The aims of this study are to 1) develop a protocol-based, promotora-led lifestyle intervention (PLI) to promote weight loss in at-risk Latinas, and assess its feasibility; 2) compare changes in weight and cardiometabolic markers-hemoglobin A1C, fasting lipids, blood pressure-from baseline to 1 year between at-risk Latinas randomly assigned to the PLI group versus metformin and usual care (UC) groups; and 3) understand the social and cultural context surrounding weight-related behaviors among Latinas at-risk for diabetes. The investigators hypothesize that Latinas assigned to PLI and metformin will have greater weight loss (primary outcome) and greater improvements in cardiometabolic markers from baseline to 1 year than those randomized to UC

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Latino ethnicity
* Spanish fluency
* Age ≥20 years
* BMI ≥25 kg/m2
* And "increased risk of diabetes" (ADA Diabetes Risk Score ≥4 as determine by 7-item questionnaire and hemoglobin A1C ≥ 5.6%)

Exclusion Criteria:

* Hemoglobin A1C ≥ 6.5%
* Current or planned pregnancy during the study period
* Chronic conditions that could affect potential participants' ability to participate (osteoarthritis, heart disease, pulmonary disease requiring oxygen or daily bronchodilator use, and severe psychiatric disease)
* Medical comorbidities that could influence weight loss or weight gain (thyroid disease, cancer, and HIV)
* Medications that could affect weight or glucose metabolism (thiazide diuretics, β-blockers, and systemic glucocorticoids).

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, MD, MSc, Principal Investigator — Temple University
Locations (1):
- Temple University - Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Promotora-led Intervention: The PLI consists of a core curriculum or 12 group sessions of 90 minute duration over a 12-week period and will be followed by a maintenance phase of 10 biweekly and then monthly 90-minute sessions during months 4 through 12. One promotora will lead each session in Spanish, exploring such topics as being active, low-fat diets, portion control, self monitoring, problem solving and life-style changes.
  Prometra led intervention: Behavioral life-style program lead by a team of trained community health workers (called promotoras) with 2 principal goals - encouraging participants to lose 7% of their total weight and complete 150 minutes of moderate physical activity per week.
Period: Overall Study
Arm/Group | Promotora-led Intervention | Usual Care | Metformin Therapy
Started | 33 | 30 | 29
Completed | 30 | 28 | 27
Not Completed | 3 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Pregnancy | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promotora-led Intervention | Usual Care | Metformin Therapy | Total
Number analyzed (Participants) | 33 | 30 | 29 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 30 | 29 | 92
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.3) | 44 (13.6) | 45.8 (11.7) | 45.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 29 | 92
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 29 | 92

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Study tests difference in body weight (Weight in kg) between treatment conditions and usual care at 12 months.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Promotora-led Intervention | Usual Care | Metformin Therapy
Number analyzed (Participants) | 30 | 28 | 27
kg | -4.0 [-5.5 to -2.6] | .8 [-.8 to 2.3] | -.9 [-2.4 to .6]

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no adverse events reported among participants.
Arm/Group | Promotora-led Intervention | Usual Care | Metformin Therapy
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/33 | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
The study was underpowered to detect a clinically meaningful weight difference between the metformin and standard care arms.

This study was a community-based translation trial with fewer eligibility criteria than DPP, a less intensive screening process, and no run-in period.

The study enrolled motivated study volunteers, potentially limiting the external validity of the findings among all Latinas with prediabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No